CLINICAL TRIAL: NCT04319731
Title: A Pilot Study of Human Amniotic Fluid for COVID19 Associated Respiratory Failure
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 131618
Record Dates: First submitted 2020-03-22; First posted 2020-03-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2020-04

CONDITIONS: SARS CoV-2 Infection
Keywords: Amniotic fluid; Respiratory failure; Critical illness
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency; Critical Illness | interventions — amniotic fluid peptide-1, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): Treatment groups:
  1. Acute care and ICU - 10mL intravenous amniotic fluid every 24 hours for 5 days (6mL)
  Interventions: Biological: Human Amniotic Fluid

INTERVENTIONS:
Biological: Human Amniotic Fluid — Administration of amniotic fluid in SARS-CoV-2 positive patients

SUMMARY:
The purpose of this study is to test the effect of purified (acellular) amniotic fluid as a treatment for SARS CoV-2 (COVID19)-associated respiratory failure. Past use of human amniotic products (i.e., membrane and fluid) is FDA-approved for tissue injury and has been used to reduce inflammation and fibrosis in patients with a variety of medical conditions. The investigators hypothesize that using nebulized and/or intravenous purified (acellular) amniotic fluid will reduce both inflammation in patients hospitalized for in SARS CoV-2 (COVID19)-associated respiratory failure, potentially leading to a decrease in respiratory support.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18
* 2. Hospitalized and symptomatic (cough, fevers, SOB, or sputum production)
* 3. SARS CoV-2 laboratory positive obtained within 14 days of enrollment

Exclusion Criteria:

* 1. None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Ventilator Free Days | Measured from hospital admission day 60 after admission.
  Days alive and off mechanical ventilation at day 60. Measured only among patients who receive invasive mechanical ventilation.
Duration of supplemental oxygen use | Measured from hospital admission to day 60.
  Duration from hospital admission until cessation of supplemental oxygen use. Measured only among patients who do not receive invasive mechanical ventilation.

SECONDARY OUTCOMES:
All cause mortality | Measured at day 60 or at hospital discharge, whichever comes first.
  Survival at day 60 or hospital discharge
Systemic inflammation | Measured at day 5 post enrollment.
  Systemic inflammation at 5 days measured by serum IL-6.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Selzman, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Health, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Selzman CH, Tonna JE, Pierce J, Vargas C, Skidmore C, Lewis G, Hatton ND, Phillips JD. A pilot trial of human amniotic fluid for the treatment of COVID-19. BMC Res Notes. 2021 Jan 22;14(1):32. doi: 10.1186/s13104-021-05443-9. PMID 33482902